CLINICAL TRIAL: NCT01649960
Title: Role of Exercise and Low-Dose Rapamycin on Age-Associated Impairments in Older Adults With Coronary Artery Disease: Cardiac Rehabilitation And Rapamycin in Elderly (CARE) Trial
Brief Title: Exercise and Low-Dose Rapamycin in Older Adults With CAD:Cardiac Rehabilitation And Rapamycin in Elderly (CARE) Trial
Acronym: CARE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-007896
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Aging; CAD
Keywords: Aging; Biomarkers; CAD
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapamycin (Other): Oral rapamycin was given during the nonrandomized phase of the study. The doses that were used of rapamycin were 0.5mg, 1mg, or 2mg.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Oral tablets were given in the dose of 0.5mg, 1mg, or 2mg once a day. This was a pilot study and the serum rapamycin levels were kept below 6ng/ml.

SUMMARY:
The investigators will do the study in two phases. The first phase will be a pilot study on up to 18 participants [patients 60 years or older with coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG) or patients who are eligible to undergo and participate in cardiac rehabilitation (CR)]; up to 6 participants each will be given oral daily rapamycin (0.5, 1, and 2mg) dose for the duration of CR. Baseline and follow-up data will be collected for age-associated impairment (AAI): frailty (primary endpoint) and quality of life (QOL),senescent-associated secretory phenotype (SASP)and abdominal/thigh subcutaneous adipose biopsy for measurement of adipocyte mitochondrial DNA copy number and to quantitate the number of senescent preadipocytes. Safety of rapamycin will be assessed by periodic clinical follow-up, blood draws, and serum rapamycin levels. Following completion of the pilot phase, the data will be analyzed. If favorable changes are noted in the SASP or AAI, the investigators will start a phase 2 randomized trial.

Second phase: In a prospective, randomized, clinical trial design, patients 60 years or older will be randomized at the time of CR to a standardized exercise protocol, or exercise protocol with the addition of low-dose rapamycin to test the hypothesis whether low-dose rapamycin (demonstrated in the pilot trial to improve SASP/AAI) will improve measures of AAI, SASP, or findings on the fat biopsy as compared to exercise alone. The null hypotheses are that there is no improvement with rapamycin in measures of AAI or SASP.

DETAILED DESCRIPTION:
Participants:

Pilot study: Patients, 60 years or older, selected for this single-center open label pilot study will be consented for participation at initiation of CR following PCI or CABG. We will enroll up to 18 patients; no more than 6 patients will receive a dose at one of the three proposed levels:0.5mg, 1.0mg, and 2mg daily oral rapamycin for the duration of CR (typically 12 weeks). We will perform physical performance tests for frailty assessment, short-form 12 for quality of life, and tests for SASP [(IL-6), matrix metalloproteinase (MMP) 3, and monocyte chemotactic protein (MCP) 1], and abdominal/thigh subcutaneous adipose biopsy for measurement of adipocyte mitochondrial DNA copy number and to quantitate the number of senescent preadipocytes. at baseline and at the conclusion of CR. Fasting lipid panel will be performed at baseline and at the completion of CR. Baseline complete blood count, liver, and kidney functions will be performed. These tests will be repeated at 14 days, 30 days, 8 weeks, and at the completion of CR. Serum rapamycin levels will be measured at 7, 14, 30 days, and at the completion of CR. The serum levels of the drug will be kept below 6ng/ml. If the drug levels were found to be higher, next low dose of the medication will be prescribed. Participants with serious side effects (appendix) from the medications will be withdrawn from the study.

Patients will be enrolled in sets of three. Thirty days of monitoring must pass on all three subjects before three more may be enrolled. The first three patients will be assigned to the 0.5 mg dose level. If two patients of those three have serious adverse events, the pilot study will be terminated. If 1 of 3 patients has an serious adverse event, we will enroll three more subjects at the 0.5 mg level. If those three have no serious events or if there were no events in the first three subjects, then we will proceed to enroll three subjects at the 1.0mg level. Otherwise, if there are 2 or more serious events in the 6 patients assigned to 0.5mg, we will terminate the study. We will proceed similarly with the 1.0 mg level before enrolling patients to the 2.0 mg level. If we observe 2 serious events at the 1.0 mg level and only 3 patients have been enrolled at the 0.5mg level, we will finish the pilot by enrolling 3 more at the 0.5 mg level. Similarly, if we observe 2 serious events at the 2.0 mg level and only have 3 subjects (with 0 events) at the 1.0 level, we will enroll 3 more at the 1.0 level.

Randomized Trial: The Cardiac rehabilitation And Rapamycin in Elderly (CARE) study is a prospective, randomized, phase 2 clinical trial that will be done at Mayo Clinic, Rochester, MN. The pool of potential study participants will consist of all patients 60 years or older with CAD who are referred to the CR following PCI or CABG. To minimize the drop out rate, we will obtain consent at the end of first week of CR participation, since most patients who quit CR do so in the first week. Consent will be obtained by the study coordinator.

Baseline Assessment:

Following informed consent, assessments of height, weight, and blood pressure will be made, and all participants will have a chemistry 15 panel, complete blood cell count, and an electrocardiogram. Race and ethnicity will be self-reported. Baseline demographic, angiographic, and other relevant clinical and laboratory data will be entered prospectively into a database.

Biochemical parameters: The mechanisms through which rapamycin retard cellular senescence and extend life span are still unclear. With this aim, a better understanding of effects of rapamycin on inflammation, mitochondrial DNA copy number, quantitation of senescent preadipocytes and diverse biomarkers of aging could be demonstrated. To assess the effect of CR, we will assess these parameters at baseline and then at the completion of the CR program.

SASP: Proinflammatory biomarkers, IL-6, MMP 3 and MCP 1 will be studied (ELISA).

Patients will be randomized in a 1:1 ratio to either regular CR, or CR with the addition of 0.5mg/1.0mg/2.0mg of rapamycin. The lowest dose of rapamycin that demonstrates potential to reduce SASP, and/or improve AAI in the pilot trial will be used.

Inclusion Criteria

1. Age 60 years or older
2. Patients eligible for CR.
3. Informed written consent.

Exclusion criteria

1. Class III or IV CHF.
2. Creatinine > 2.0 mg/dl.
3. HbA1c > 13%.
4. Any malignancy
5. Hematological disorder, including thrombocytopenia, leucopenia.
6. Noncardiac illness expected to limit survival.
7. Chronic liver disease.
8. Suspected or known pregnancy.
9. Geographically inaccessible or unable to return for follow-up.
10. Unable to understand or cooperate with protocol requirements.

12. Post organ transplant or with immune-compromised status 13. Prior stroke with disability, severe Parkinson disease 14. Dementia 15. Post-CABG <3 months or any evidence of active wounds or ulcers. 16.Anticipating elective surgery in the 3 months following enrollment.

ELIGIBILITY:
Inclusion Criteria

1. Age 60 years or older
2. Patients eligible to undergo cardiac rehabilitation.
3. Informed written consent.

Exclusion criteria

1. Class III or IV CHF.
2. Creatinine > 2.0 mg/dl.
3. HbA1c > 13%.
4. Any malignancy
5. Hematological disorder, including thrombocytopenia, leucopenia.
6. Noncardiac illness expected to limit survival.
7. Chronic liver disease.
8. Suspected or known pregnancy.
9. Geographically inaccessible or unable to return for follow-up.
10. Unable to understand or cooperate with protocol requirements.
11. Post organ transplant or with immune-compromised status
12. Prior stroke with disability, severe Parkinson disease
13. Dementia
14. Post-CABG <3 months or any evidence of active wounds or ulcers.
15. Anticipating elective surgery in the 3 months following enrollment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frailty | Twelve months
  Frailty will be measured using physical performance tests, gait speed, and grip strength.

SECONDARY OUTCOMES:
Senescent-associated secretory phenotype | twelve months
  The SASP will include interleukin 6, Matrix metalloproteinase 3, and Monocyte chemotactic protein 1.

OTHER OUTCOMES:
Quality of life | Twelve months
  Short-form 12 will be measured
Mitochondrial DNA copy number and quantitation of senescent preadipocytes | 12 weeks, before and after cardiac rehabilitation
  These variables will be analyzed by a fat biopsy (abdominal/thigh) before and following completion of cardiac rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester and Mayo Health System sites in Austin and Albert Lea, Minnesota, Rochester, Minnesota, United States

REFERENCES:
- [Result] Singh M, Jensen MD, Lerman A, Kushwaha S, Rihal CS, Gersh BJ, Behfar A, Tchkonia T, Thomas RJ, Lennon RJ, Keenan LR, Moore AG, Kirkland JL. Effect of Low-Dose Rapamycin on Senescence Markers and Physical Functioning in Older Adults with Coronary Artery Disease: Results of a Pilot Study. J Frailty Aging. 2016;5(4):204-207. doi: 10.14283/jfa.2016.112. PMID 27883166